CLINICAL TRIAL: NCT02438254
Title: Oklahoma Family Health Patterns: A Study Across Generations
Brief Title: Texas Family Health Patterns: A Study Across Generations
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 14-410H; 2R01AA012207-11 (NIH)
Record Dates: First submitted 2015-04-23; First posted 2015-05-08 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Alcohol and Other Drug Use Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FH+: Young adults with at least one parent with an alcohol or other drug use disorder history.
- FH-: Young adults with no histories of alcohol or other drug use disorders in any parents or grandparents.

SUMMARY:
The researchers are studying factors that may increase the risk for alcohol and drug use in individuals who do not have any problems with these substances. This study will be looking at health behaviors in young adults compared to their family's health behaviors and lifestyle.

The investigators plan to study genetic differences in people with and without a family history of alcoholism. The researchers hope to learn how a family history of alcoholism, early life adversity and different genotypes shape personal characteristics associated with a risk for alcoholism.

DETAILED DESCRIPTION:
The Oklahoma Family Health Patterns project is an intensive study of psychological, behavioral, and stress reactivity characteristics in healthy young adults with a family history of alcoholism (FH+) with a goal of identifying characteristics that place these persons at elevated risk for the disorder. The investigators have recently identified early life adverse experience (ELA), including physical and sexual abuse and separation from parents, as occurring with disproportionate impact in FH+, and the investigators have shown that ELA accounts for diminished stress reactivity, behavioral impulsivity, and poor mood regulation, all of which are risk factors for alcohol and other substance use disorders. The impact of ELA in the FH+ population demands to be studied further in a Gene x Environment interaction given the known positive feedbacks between FH+ and ELA. The investigators' goal is to carry out a G x E interaction study by genotyping the investigators' FH x ELA and examining the impact of genotype on the broad range of personal characteristics currently under study in this project. Aim 1. Examine the differential impact of ELA on psychological and behavioral characteristics of FH+ vs. FH- groups using an expanded sample of volunteers. Aim 2. Use the investigators' larger sample to carry out a Gene x Environment analysis to test specific alleles that are strongly suspected of influencing activity in brain motivational systems, expanding on work the investigators initiated with NIAAA thanks to a supplement to this R01 (AA012207-S1). Aim 3. Test specific aspects of temperament as endophenotypes linking FH and ELA to behavioral, cognitive, and stress reactivity as aspects of the person's phenotype. Aim 4. Increase the investigators' recruitment base by screening and testing volunteers at a second site, the University of Texas HSC, San Antonio, where the investigators currently conduct our neuroimaging studies. Alcoholism is a costly burden to society, but risk factors for alcoholism are poorly understood. The vast majorities of studies focuses on alcoholic patients but are unable to disentangle preexisting influences from the effects of alcohol intake history. The investigators' high-risk study design can be of value by contrasting FH+ and FH- with regard to environmental contributors and genetic vulnerabilities that contribute to behavioral risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Male or female sex
* Age 18-29 years
* Normal health based on routine history and physical
* Willingness to provide a DNA sample
* No required CNS-acting medications, history of neurological impairment, or diabetes mellitus
* Normal color vision
* Normal intelligence based on Shipley Institute of Living verbal scale score ≥ 20 (John & Rattan, 1992)
* Negative urine drug screen at entry and each lab visit (icup, Alcopro, Knoxville, TN) and alcohol breath test (AlcoMate CA2000, KHN Solutions, San Francisco)
* Volunteers must have been raised by at least one biological parent and have knowledge of and contact with same

Exclusion Criteria:

* Pregnancy
* Any failure to meet inclusion criteria
* Rearing by other than a biological parent
* Suspected maternal alcoholism during pregnancy with proband, determined by interview with subject or parent
* AUDIT score > 12
* Inability of parent to provide credible report of family alcohol use patterns for two generations
* Current Axis I disorder by DIS-IV, excepting past depression or abuse of alcohol or drugs (all > 60 days)
* Axis II disorder in Clusters A or C by SCID II. AXIS II symptoms in Cluster B are not exclusionary because antisocial and behavioral undercontrol variables related to substance use disorders overlap with Cluster B symptoms. Past abuse of alcohol and other substances is not exclusionary in order to allow a wide range of intake while still avoiding severe consequences of intake history.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young adults with at least one parent with an alcohol or other drug use disorder history (FH+) or no alcohol or other drug use disorders in any parents or grandparents (FH-).
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Assess behavioral risk factors in young adults with and without family histories of alcohol and other drug use disorders | Participants will be assessed on 3 laboratory visits lasting a few hours each. All 3 visits will typically be competed within 3-4 weeks.
Collect physiological measures of stress reactivity in young adults with and without family histories of alcohol and other drug use disorders | Participants will be assessed on 3 laboratory visits lasting a few hours each. All 3 visits will typically be competed within 3-4 weeks.
Collect DNA in young adults with and without family histories of alcohol and other drug use disorders | DNA will be collected once during one of the participants' 3 laboratory visits lasting a few hours each. All 3 visits will typically be competed within 3-4 weeks. .
Maintain DNA repository for DNA analyses | The DNA repository will be maintained over the 5 year study duration.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States